CLINICAL TRIAL: NCT02718339
Title: In-patient Asthma Counseling by Pulmonologist and Hospital Re-admission Rate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SOR-169-15 CTIL
Record Dates: First submitted 2016-03-20; First posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive counseling by a pulmonologist (Experimental): Counselor visit during hospitalization, telephone follow up for 4 weeks and a follow up visits.
  Interventions: Behavioral: Intensive counseling
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Intensive counseling
  Arms: Intensive counseling by a pulmonologist

SUMMARY:
Prospective randomized clinical trial to assess the effect of in-hospital intensive counseling and follow-up vs. usual care, on re-admission rates of patients with Asthma.

The study population will include asthma patients admitted to internal Medicine departments and medical ICU at Soroka University Medical Center, due to asthma exacerbation.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years old.
2. Admitted to Internal Medicine at Soroka University Medical Center due to asthma exacerbation.

Exclusion Criteria:

1. Substance abuse (except for tobacco).
2. Handicapped or bed ridden patients.
3. Patients who don't speak Hebrew, English, Russian or Arabic.
4. Other significant respiratory disease such as COPD, interstitial lung disease (as decided by the PI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Re-admission rate | Within 6 months after discharge